CLINICAL TRIAL: NCT02567825
Title: Efficacy of Tympanostomy Tubes for Children With Recurrent Acute Otitis Media
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alejandro Hoberman (Other)
Collaborators: George Washington University (Other); National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor-Investigator, Alejandro Hoberman, Professor of Pediatrics, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRO15060148; 1U01DC013995-01A1 (NIH)
Record Dates: First submitted 2015-10-01; First posted 2015-10-05 (Estimated); Results first posted 2021-12-10 (Actual); Last update posted 2022-07-15 (Actual); Status verified 2022-06

CONDITIONS: Acute Otitis Media
Keywords: ear infection; antibiotics; infants; children; pediatrics; tympanostomy tubes
MeSH Terms: conditions — Otitis Media; Otitis

STUDY DESIGN:
Masking Description: Subjects in the randomization phase of the study will be randomized to either medical management or tube surgery. No masking will occur.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Surgical Management (Active Comparator): Tympanostomy Tube Placement Topical antimicrobial treatment of acute otitis media episodes with ofloxacin drops
  Interventions: Device: Tympanostomy tube placement; Drug: Ofloxacin Otic
- Non-Surgical Management (Other): Antimicrobial treatment of acute otitis media episodes with amoxicillin-clavulanate and/or ceftriaxone
  Interventions: Drug: Amoxicillin-Clavulanate and/or Ceftriaxone

INTERVENTIONS:
Device: Tympanostomy tube placement — As per routine care, tympanostomy tubes will be inserted under general anesthesia, using a small radial incision in the anteroinferior portion of the tympanic membrane; a Teflon® Armstrong-type tympanostomy tube will be used.
  Arms: Surgical Management
Drug: Amoxicillin-Clavulanate and/or Ceftriaxone — Children randomized to nonsurgical management will receive stepwise therapy with amoxicillin-clavulanate (90/6.4 mg/kg in two divided doses for 10 days), and in the event of inadequate response, ceftriaxone (75 mg/kg intramuscularly, repeated in 48 hours), as recommended in the American Academy of Pediatrics guidelines.
  Arms: Non-Surgical Management
Drug: Ofloxacin Otic — Participants randomized to receive tympanostomy tubes will also be followed overtime for recurrences of AOM and treated with topical ofloxacin (Floxin® 0.3%, 5 mL) 5 drops into the affected ear twice daily for 10 days. Persistence of otorrhea after 7 days of treatment will be considered inadequate response, and children so affected will be prescribed empiric amoxicillin-clavulanate (90/6.4 mg/kg/day in two divided doses) followed by culture-directed therapy 48 hours later.
  Arms: Surgical Management

SUMMARY:
To determine whether tympanostomy tube placement (TTP) compared with nonsurgical management will meaningfully improve children's acute otitis media (AOM) experience over the succeeding 2 years.

DETAILED DESCRIPTION:
Tympanostomy tube placement (TTP) for recurrent acute otitis media (rAOM) is frequently performed in children under 3 years of age; however, a critical need exists to establish its risk/benefit ratio. Seventy percent of children experience at least one episode of AOM during the first year of life; 20% of children have rAOM. The efficacy of TTP for preventing rAOM, assumedly by maintaining middle-ear ventilation, remains unclear. Benefits of TTP must be balanced against risks of anesthesia, complications and sequelae of surgery, and cost. Accordingly, the objective of this proposal is to determine the efficacy of TTP in children aged 6-35 months, the group in which rAOM is most troublesome. The central hypothesis is that in children with rAOM, the operation will prove effective over the ensuing 2 years overall, but the benefit in a more severely affected, and therefore higher-risk subgroup may be substantially greater than in a less severely affected subgroup, in whom benefits may not outweigh risks. The rationale for this research is based on a belief that the limited nature of the benefit of TTP found in earlier clinical trials may have been the result of enrolling children whose illnesses had not been diagnosed using stringent criteria and/or whose ascertainment of episodes had relied on undocumented histories. The primary objective is to determine the extent to which TTP reduces the overall rate of recurrences in children with rAOM over a 2-year period. In a randomized, clinical trial, children aged 6-35 months who are at risk for rAOM will be followed prospectively and examined promptly with new respiratory illnesses to accurately document episodes of AOM. A total of 240 children who meet stringent inclusion criteria for rAOM will be eligible to undergo randomization within strata (age and exposure to other children) to receive TTP or nonsurgical management. Children will be followed for 2 years; the average number of episodes of AOM will be documented and compared between groups. The secondary objective is to determine changes following TTP in nasopharyngeal (NP) colonization with resistant bacteria. At the time of randomization and 3 times a year for 2 years, NP specimens will be obtained and cultured. Susceptibility testing and serotyping will be performed, and the proportions of children colonized with resistant bacteria compared between treatment groups. The tertiary objective is to determine cost-effectiveness of TTP. The investigators will calculate both direct medical and nonmedical costs and correlate this with the number of days that each child has AOM symptoms, otorrhea, and any adverse events or complications. The proposed research is innovative, as the investigators will document AOM episodes prospectively using stringent diagnostic criteria and obtain digital tympanic membrane images otoendoscopically to enhance accuracy of observations. Findings of the proposed study will provide clinicians and parents with dependable evidence concerning the overall effects of TTP compared with nonsurgical management in children with rAOM of varying degrees of severity, enabling evidence-based decisions regarding an important component of the children's healthcare.

ELIGIBILITY:
Inclusion Criteria

1. are aged 6-35 months,
2. have rAOM, defined as the occurrence of 3 AOM episodes in 6 months or 4 episodes in 12 months with ≥1 episode in the preceding 6 months, and
3. 2 of these AOM episodes have been documented by trained study personnel.

Exclusion Criteria

1. have a history of TTP,
2. have a chronic illness (cystic fibrosis, neoplasm, juvenile diabetes, renal or hepatic insufficiency, immune dysfunction, malabsorption, inflammatory bowel disease, severe asthma requiring at least 4 courses of oral corticosteroids during the last 12 months),
3. are allergic to amoxicillin,
4. have a congenital anomaly that might increase the risk of recurrences (e.g., cleft palate, Down's syndrome),
5. have had otitis media effusion for at least 3 months in addition to rAOM, or
6. have sensorineural hearing loss.

Ages: 6 Months to 35 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 250 (Actual)
Dates: Start 2015-11; Primary Completion 2020-03 (Actual); Study Completion 2021-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alejandro Hoberman, MD, Principal Investigator — University of Pittsburgh School of Medicine; Children's Hospital of Pittsburgh of UPMC; Diego Preciado, MD, PhD, Principal Investigator — George Washington University; Childrens National Medical Center
Locations (2):
- United States (2):
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Noorbakhsh KA, Liu H, Kurs-Lasky M, Smith KJ, Hoberman A, Shaikh N. Cost-Effectiveness of Management Strategies in Recurrent Acute Otitis Media. J Pediatr. 2023 May;256:11-17.e2. doi: 10.1016/j.jpeds.2022.11.032. Epub 2022 Dec 5. PMID 36470464
- [Derived] Hoberman A, Preciado D, Paradise JL, Chi DH, Haralam M, Block SL, Kearney DH, Bhatnagar S, Muniz Pujalt GB, Shope TR, Martin JM, Felten DE, Kurs-Lasky M, Liu H, Yahner K, Jeong JH, Cohen NL, Czervionke B, Nagg JP, Dohar JE, Shaikh N. Tympanostomy Tubes or Medical Management for Recurrent Acute Otitis Media. N Engl J Med. 2021 May 13;384(19):1789-1799. doi: 10.1056/NEJMoa2027278. PMID 33979487

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Surgical Management | Non-Surgical Management
Started | 129 | 121
Completed | 108 | 100
Not Completed | 21 | 21
Not completed — No follow-up post-randomization | 5 | 1
Not completed — Follow-up less than 23 months | 16 | 20

BASELINE CHARACTERISTICS:
Population: 250 children underwent randomization; 129 were randomized to surgical management and 121 to non-surgical management. The 129 and 121 participants, respectively, were the basis for analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Surgical Management | Non-Surgical Management | Total
Number analyzed (Participants) | 129 | 121 | 250
Age, Customized [Count of Participants; unit: Participants]
  6-11 months | 46 | 45 | 91
  12-23 months | 70 | 67 | 137
  24-35 months | 13 | 9 | 22
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 48 | 90
  Male | 87 | 73 | 160
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Ethnicity was reported by the parent.
  Participants
    Hispanic or Latino | 19 | 10 | 29
    Not Hispanic or Latino | 110 | 111 | 221
    Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Race was reported by the parent.
  Participants
    American Indian or Alaska Native | 1 | 0 | 1
    Asian | 3 | 2 | 5
    Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
    Black or African American | 41 | 42 | 83
    White | 70 | 70 | 140
    More than one race | 10 | 7 | 17
    Unknown or Not Reported | 3 | 0 | 3
Site of Enrollment [Count of Participants; unit: Participants] — Measure Description: Participating clinical study sites included: Children's Hospital of Pittsburgh (CHP) of University of Pittsburgh Medical Center (UPMC), Pittsburgh, Pennsylvania; Children's National Medical Center (CNMC), Washington, District of Columbia; and Kentucky Pediatric/Adult Research (KPAR) and Physicians to Children and Adolescents (PTCA) Bardstown, Kentucky.
  Participants
    Children's Hospital of Pittsburgh (CHP) | 92 | 91 | 183
    Children's National Medical Center (CNMC) | 20 | 16 | 36
    Kentucky Pediatric and Adult Research (KPAR) | 17 | 14 | 31
Maternal Level of Education [Count of Participants; unit: Participants] — Parent was asked about the highest level of maternal education. High school graduate or equivalent implies the mother has graduated high school, or has a General Education Diploma (GED), or has attended technical school or some college, or has an associates degree.
  Participants
    Less than high school | 6 | 4 | 10
    High school graduate or equivalent | 62 | 55 | 117
    College graduate | 52 | 56 | 108
    Unknown | 9 | 6 | 15
Type of Health Insurance [Count of Participants; unit: Participants] — Type of health insurance relates to the child's insurance.
  Participants
    Private | 62 | 62 | 124
    Public | 63 | 59 | 122
    None | 4 | 0 | 4
Exposure to Other Children [Count of Participants; unit: Participants] — Exposure to other children was defined as exposure to at least 3 children for at least 10 hours per week.
  Participants
    No | 26 | 22 | 48
    Yes | 103 | 99 | 202
Otitis Media With Effusion (OME) Present at Randomization [Count of Participants; unit: Participants]
  No | 85 | 71 | 156
  Yes | 44 | 50 | 94
Estimated Risk of Recurrences of Acute Otitis Media (AOM) [Count of Participants; unit: Participants] — Risk of recurrences was based on early age of onset of AOM; numerous and/or frequent previous AOM episodes; receipt of multiple courses of antibiotic; eligibility for enrollment first evident during warm-weather months; parental characterization of previous AOM episodes as severe; eligibility for enrollment despite nonexposure to other young children; moderate or marked tympanic membrane (TM) bulging with previous AOM episodes; most previous AOM episodes in both ears; and a high score on the Acute Otitis Media Severity of Symptom scale during screening and/or at enrollment.
  Participants
    Low risk | 63 | 72 | 135
    High risk | 66 | 49 | 115

OUTCOME MEASURES:

1. Primary Outcome: The Rate of Occurrence of Acute Otitis Media (AOM) Episodes Per Child-Year
Description: An episode of AOM is considered a discrete occurrence if symptoms and signs persisted for, or recurred, 17 or more days after the start of antimicrobial treatment. The rate is calculated by dividing the total number of occurrences by the total number of years of follow-up. Multiple imputation was used when follow-up was incomplete.
Time Frame: Day 1 until Day 786. The mean length of actual follow-up was 662 days / 1.8 years. For each child with incomplete 2-year follow-up, multiple imputation was used and values for the remaining days/years were imputed.
Population: The analysis was intention-to-treat (ITT). The participants are randomized children. For each child with incomplete 2-year follow-up, the total number of episodes of acute otitis media were imputed using multivariate imputation by chained equations with 50 imputations.
Measure: Mean (Standard Error); unit: Occurrences per child-year
Arm/Group | Surgical Management | Non-Surgical Management
Number analyzed (Participants) | 129 | 121
Occurrences per child-year | 1.48 (.08) | 1.56 (.08)
Statistical Analysis 1: Comparison: Surgical Management vs Non-Surgical Management; Null hypothesis: There is no difference between the two groups in the rate of occurrence of AOM per child-year during the 2-year follow-up period; Test type: Superiority; p = 0.66, Generalized linear model; The p-value is adjusted for site, age at enrollment, and exposure or nonexposure to other children; Risk Ratio (RR) = 0.97, 95% CI 2-sided [0.84 to 1.12] — The Surgical Management group represents the numerator for the risk ratio and the Non-Surgical Management group represents the denominator. The estimates are adjusted for site, age at enrollment, and exposure or nonexposure to other children

2. Secondary Outcome: The Rate of Occurrence of Acute Otitis Media (AOM) Episodes Per Child-Year According to the Estimated Risk of Acute Otitis Media (AOM) Recurrences at Enrollment
Description: An episode of AOM is considered a discrete occurrence if symptoms and signs persisted for, or recurred, >=17 days after the start of antimicrobial treatment. The rate is calculated by dividing the total # of occurrences by the total # of years of follow-up. Risk of recurrences was based on early age of onset of AOM; numerous and/or frequent previous AOM episodes; receipt of multiple courses of antibiotic; eligibility for enrollment first evident during warm-weather months; parental characterization of previous AOM episodes as severe; eligibility for enrollment despite nonexposure to other young children; moderate or marked tympanic membrane (TM) bulging with previous AOM episodes; most previous AOM episodes in both ears; and a high score on the Acute Otitis Media Severity of Symptom scale (with scores ranging from 0 to 10 and higher scores indicating greater severity of symptoms) during screening and/or at enrollment. Multiple imputation was used when follow-up was incomplete.
Time Frame: as for outcome 1
Population: The analysis was ITT. The participants are randomized children. For each child with incomplete 2-year follow-up, the total number of episodes of acute otitis media were imputed using multivariate imputation by chained equations with 50 imputations.
Measure: Mean (Standard Error); unit: Occurrences per child-year
Arm/Group | Surgical Management | Non-Surgical Management
Number analyzed (Participants) | 129 | 121
Occurrences per child-year
  Children considered at low risk of AOM recurrence: number analyzed (Participants) | 63 | 72
  Children considered at low risk of AOM recurrence | 1.28 (0.10) | 1.56 (0.10)
  Children considered at high risk of AOM recurrence: number analyzed (Participants) | 66 | 49
  Children considered at high risk of AOM recurrence | 1.67 (0.11) | 1.56 (0.13)
Statistical Analysis 1: Comparison: Surgical Management vs Non-Surgical Management; Null hypothesis: There is no difference between the two groups in the rate of occurrence of AOM per child-year during the 2 year follow-up among children considered at low risk of AOM recurrences at enrollment; Test type: Superiority; Risk Ratio (RR) = 0.82, 95% CI 2-sided [0.67 to 1.01] — The Surgical Management group represents the numerator for the risk ratio and the Non-Surgical Management group represents the denominator
Statistical Analysis 2: Comparison: Surgical Management vs Non-Surgical Management; Null hypothesis: There is no difference between the two groups in the rate of occurrence of AOM per child-year during the 2 year follow-up among children considered at high risk of AOM recurrences at enrollment; Test type: Superiority; Risk Ratio (RR) = 1.07, 95% CI 2-sided [0.86 to 1.33] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: Surgical Management vs Non-Surgical Management; Null hypothesis: There is no interaction between comparison group (Surgical Management, Non-Surgical Management) and risk group (children considered at low risk of AOM recurrences at enrollment, children considered at high risk of AOM recurrences at enrollment); Test type: Other; p = 0.08, Generalized linear models

3. Secondary Outcome: The Frequency Distribution of AOM Episodes Among Children Completing the Study
Description: An episode of AOM is considered a discrete occurrence if symptoms and signs persisted for, or recurred, 17 or more days after the start of antimicrobial treatment. Children with at least 23 months of follow-up were considered to have completed the study.
Time Frame: Day 1 until Day 786. For children completing the study, the mean length of follow-up was 726 days.
Population: The analysis was ITT. The participants are randomized children having follow-up greater than or equal to 23 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Surgical Management | Non-Surgical Management
Number analyzed (Participants) | 108 | 100
Participants
  Number of cumulative episodes = 0 | 17 | 12
  Number of cumulative episodes = 1 or 2 | 41 | 41
  Number of cumulative episodes = 3 or 4 | 24 | 29
  Number of cumulative episodes >= 5 | 26 | 18
Statistical Analysis 1: Comparison: Surgical Management vs Non-Surgical Management; Null hypothesis: There is no difference between the two groups in the proportion of children completing the study with 0, 1 or 2, 3 or 4, greater than or equal to 5 episodes of AOM; Test type: Superiority; p = 0.48, Chi-squared

4. Secondary Outcome: The Distribution of Children Experiencing Treatment Failure (TF)
Description: Parents used the Acute Otitis Media Severity of Symptoms (AOM-SOS) scale (version 4.0) to rate each of 5 symptoms as none, a little, or a lot, with corresponding scores of 0, 1, and 2. Total scores range from 0 to 10; higher scores indicate greater severity of symptoms. AOM episodes were categorized as likely severe if the parent described the child as having moderate or severe otalgia (a lot of ear tugging), temperature ≥39°C, or an AOM-SOS scale score >6 Day 1 of the episode. TF is defined as frequent AOM recurrences (2 in 3 months, 3 in 6 or 4 in 12); ≥3 likely severe AOM recurrences, receipt of ≥45 cumulative days of systemic antimicrobial treatment for AOM, otorrhea for ≥45 cumulative days or diarrhea associated with antimicrobial treatment for ≥30 cumulative days, respectively, in 12 months; persistent effusion for ≥12 successive months; TM perforation for ≥90 days; AOM related hospitalization; anesthesia reactions; and tubes in children randomized to nonsurgical management.
Time Frame: Day 1 until Day 786.
Population: The analysis was ITT. The participants are randomized children with follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Surgical Management | Non-Surgical Management
Number analyzed (Participants) | 124 | 120
Participants
  Experienced failure | 56 | 74
  Did not experience failure | 68 | 46
Statistical Analysis 1: Comparison: Surgical Management vs Non-Surgical Management; Null hypothesis: There is no difference between the two groups in the proportion of children experiencing treatment failure; Test type: Superiority; Risk Ratio (RR) = 0.73, 95% CI 2-sided [0.58 to 0.92] — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: The Time to the First Episode of AOM
Description: The time to the first episode of AOM is defined as the time, expressed in months, from randomization until the first episode of AOM.
Time Frame: Day 1 until Day 786. The mean length of follow-up was 662 days / 21.8 months.
Population: The analysis was ITT. The participants are randomized children.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Surgical Management | Non-Surgical Management
Number analyzed (Participants) | 129 | 121
Months | 4.34 [2.99 to 5.88] | 2.33 [1.61 to 3.12]
Statistical Analysis 1: Comparison: Surgical Management vs Non-Surgical Management; Null hypothesis: There is no difference between the two groups regarding the time to the first episode of AOM; Test type: Superiority; Hazard Ratio (HR) = 0.68, 95% CI 2-sided [0.52 to 0.90] — The Surgical Management group represents the numerator for the hazard ratio and the Non-Surgical Management group represents the denominator. The estimates are adjusted for site, age at enrollment, and exposure or nonexposure to other children

6. Secondary Outcome: The Distribution of AOM Episodes Categorized as Probably Severe or Probably Nonsevere
Description: The American Academy of Pediatrics clinical practice guideline concerning the management of AOM refers to children with "severe signs or symptoms" as those with "moderate or severe otalgia or otalgia for >= 48 hours or temperature 39°C (102.2°F) or higher." To simulate that definition, scores are used from the 5-item Acute Otitis Media Severity of Symptoms (AOM-SOS) scale (version 4.0) in which parents are asked to rate symptoms, as compared with the child's usual state, as none, a little, or a lot, with corresponding scores of 0, 1, and 2. Total scores range from 0 to 10, with higher scores indicating greater severity of symptoms. AOM episodes are categorized as "probably severe" if the parent described the child as having had moderate or severe otalgia (a lot of ear tugging; i.e. a score of 2), temperature >=39°C, or an AOM-SOS scale score >6 on Day 1 of the episode. If not "probably severe", then the episode is categorized as "probably nonsevere".
Time Frame: Day 1 until Day 786.
Population: The analysis was ITT. The participants are randomized children having at least one episode of AOM.
Measure: Count of Units; unit: Episodes of AOM
Units Other Than Participants: Episodes of AOM
Arm/Group | Surgical Management | Non-Surgical Management
Number analyzed (Participants) | 103 | 106
Number analyzed (Episodes of AOM) | 336 | 333
Episodes of AOM
  Probably nonsevere | 180 | 168
  Probably severe | 156 | 165
Statistical Analysis 1: Comparison: Surgical Management vs Non-Surgical Management; Null hypothesis: There is no difference between the two groups in the proportion of episodes categorized as probably severe; Test type: Superiority; Risk Ratio (RR) = 0.91, 95% CI 2-sided [0.76 to 1.09] — [estimate comment as in outcome 1, analysis 1]

7. Secondary Outcome: The Distribution of AOM Episodes Presenting With Tympanic Membrane Bulging or Otorrhea
Description: The presence of either tympanic membrane bulging or tympanic membrane perforation with purulent otorrhea, in addition to documentation of symptoms, is required for each episode of AOM.
Time Frame: Day 1 until Day 786.
Population: The analysis was ITT. The participants are randomized children having at least one episode of AOM.
Measure: Count of Units; unit: Episodes of AOM
Units Other Than Participants: Episodes of AOM
Arm/Group | Surgical Management | Non-Surgical Management
Number analyzed (Participants) | 103 | 106
Number analyzed (Episodes of AOM) | 336 | 333
Episodes of AOM
  Episodes presenting with tympanic membrane bulging | 86 | 248
  Episodes presenting with otorrhea | 250 | 85
Statistical Analysis 1: Comparison: Surgical Management vs Non-Surgical Management; Null hypothesis: There is no difference between the two groups in the proportion of episodes presenting with tympanic membrane bulging rather than otorrhea; Test type: Superiority; Risk Ratio (RR) = 0.34, 95% CI 2-sided [0.26 to 0.44]; The Surgical Management group represents the numerator for the risk ratio and the Non-Surgical Management group represents the denominator. The estimates are adjusted for site, age at enrollment, and exposure or nonexposure to other children

8. Secondary Outcome: The Mean Days Per Year Children Experience Tube Otorrhea
Description: Adverse events, including tube-associated otorrhea, were collected from enrollment through the end of study. Each study visit included a review of adverse events. Any such event that occurred since the previous visit was recorded, including the date of onset and the date of resolution. For each child, the days per year of tube otorrhea is calculated by dividing the total number of days of tube otorrhea (based on dates of onset and resolution) by the total number of years of follow-up.
Time Frame: Day 1 until Day 786. The mean length of follow-up was 662 days / 1.8 years.
Population: The analysis was ITT. The participants are randomized children.
Measure: Mean (Standard Error); unit: Days per year
Arm/Group | Surgical Management | Non-Surgical Management
Number analyzed (Participants) | 129 | 121
Days per year | 7.96 (1.10) | 2.83 (0.78)
Statistical Analysis 1: Comparison: Surgical Management vs Non-Surgical Management; Null hypothesis: There is no difference between the two groups in the mean days per year children experience tube otorrhea. The analysis uses a weighted regression model with weights equal to the length of follow-up; Test type: Superiority; Difference of least-squares means = 5.21, 95% CI 2-sided [2.60 to 7.82] — The Surgical Management group represents the first number in the subtraction and the Non-Surgical Management group represents the second. The estimates are adjusted for site, age at enrollment, and exposure or nonexposure to other children

9. Secondary Outcome: The Mean Days Per Year Children Experience AOM Symptoms With an Intact Tympanic Membrane (TM)
Description: For a given child, if a day of follow-up coincides with a study visit, the status of the right and left TMs are recorded at the ear exam. If a day of follow-up does not coincide with a study visit the status of each TM is assumed to be the same as the status on the prior day. Scores are used from the 5-item Acute Otitis Media Severity of Symptoms (AOM-SOS) scale (version 4.0) in which parents are asked to rate symptoms, as compared with the child's usual state, as none, a little, or a lot, with corresponding scores of 0, 1, and 2. Total scores range from 0 to 10, with higher scores indicating greater severity of symptoms. Scores are recorded at study visits and on diaries. The total number of days with an intact TM and a AOM-SOS score greater than or equal to 1 is divided by the total number of years of follow-up to arrive at the days per year with AOM symptoms and an intact TM.
Time Frame: Day 1 until Day 786. The mean length of follow-up was 662 days / 1.8 years.
Population: The analysis was ITT. The participants are randomized children.
Measure: Mean (Standard Error); unit: Days per year
Arm/Group | Surgical Management | Non-Surgical Management
Number analyzed (Participants) | 129 | 121
Days per year | 2.00 (0.29) | 8.33 (0.59)
Statistical Analysis 1: Comparison: Surgical Management vs Non-Surgical Management; Null hypothesis: There is no difference between the two groups in the mean days per year children experience AOM symptoms with an intact TM. The analysis uses a weighted regression model with weights equal to the length of follow-up; Test type: Superiority; Difference of least-squares means = -6.32, 95% CI 2-sided [-7.55 to -5.10] — [estimate comment as in outcome 8, analysis 1]

10. Secondary Outcome: The Mean Days Per Year Children Receive Systemic Antimicrobials for AOM
Description: Systemic antibiotics include Amoxicillin-Clavulanate, Ceftriaxone, Cefdinir, Amoxicillin, Azithromycin, Clindamycin, Levofloxacin, Bactrim, Cefprozil, Omnicef and Trimethoprim-Sulfamethoxazole. The days per year, for each child, is calculated by dividing the total number of days the child receives systemic antimicrobials for AOM (based on the recorded start and stop dates) by the total number of years of follow-up.
Time Frame: Day 1 until Day 786. The mean length of follow-up was 662 days / 1.8 years.
Population: The analysis was ITT. The participants are randomized children.
Measure: Mean (Standard Error); unit: Days per year
Arm/Group | Surgical Management | Non-Surgical Management
Number analyzed (Participants) | 129 | 121
Days per year | 8.76 (0.94) | 12.92 (0.90)
Statistical Analysis 1: Comparison: Surgical Management vs Non-Surgical Management; Null hypothesis: There is no difference between the two groups in the mean days per year children receive systemic antimicrobials for AOM. The analysis uses a weighted regression model with weights equal to the length of follow-up; Test type: Superiority; Difference of least-squares means = -4.50, 95% CI 2-sided [-6.82 to -2.18] — [estimate comment as in outcome 8, analysis 1]

11. Secondary Outcome: The Distribution of Children for Whom Protocol-Defined Diarrhea (PDD) Was Reported
Description: PDD is defined as the occurrence of three or more watery stools on 1 day or two or more watery stools on each of 2 consecutive days. Adverse events, including PDD, were collected from enrollment through the end of study. Each study visit included a review of medication-related adverse events. Any such event that occurred since the previous visit was recorded.
Time Frame: Day 1 until Day 786.
Population: The analysis was intention-to-treat (ITT). The participants are randomized children.
Measure: Count of Participants; unit: Participants
Arm/Group | Surgical Management | Non-Surgical Management
Number analyzed (Participants) | 129 | 121
Participants
  PDD was reported | 21 | 34
  PDD was not reported | 108 | 87
Statistical Analysis 1: Comparison: Surgical Management vs Non-Surgical Management; Null hypothesis: There is no difference between the two groups regarding the proportion of children for whom PDD was reported; Test type: Superiority; Risk Ratio (RR) = 0.67, 95% CI 2-sided [0.44 to 1.03] — [estimate comment as in outcome 5, analysis 1]

12. Secondary Outcome: The Distribution of Children for Whom Diaper Dermatitis Was Reported
Description: Diaper dermatitis is defined as diaper rash necessitating administration of topical antifungal therapy. Adverse events, including diaper dermatitis, were collected from enrollment through the end of study. Each study visit included a review of medication-related adverse events. Any such event that occurred since the previous visit was recorded.
Time Frame: Day 1 until Day 786.
Population: The analysis was ITT. The participants are randomized children.
Measure: Count of Participants; unit: Participants
Arm/Group | Surgical Management | Non-Surgical Management
Number analyzed (Participants) | 129 | 121
Participants
  Diaper dermatitis was reported | 25 | 33
  Diaper dermatitis was not reported | 104 | 88
Statistical Analysis 1: Comparison: Surgical Management vs Non-Surgical Management; Null hypothesis: There is no difference between the two groups regarding the proportion of children for whom diaper dermatitis was reported; Test type: Superiority; Risk Ratio (RR) = 0.79, 95% CI 2-sided [0.51 to 1.22] — [estimate comment as in outcome 1, analysis 1]

13. Secondary Outcome: The Distribution of Children for Whom Tube Otorrhea Was Reported
Description: Adverse events, including tube-associated otorrhea, were collected from enrollment through the end of study. Each study visit included a review of adverse events. Any such event that occurred since the previous visit was recorded.
Time Frame: Day 1 until Day 786.
Population: The analysis was ITT. The participants are randomized children.
Measure: Count of Participants; unit: Participants
Arm/Group | Surgical Management | Non-Surgical Management
Number analyzed (Participants) | 129 | 121
Participants
  Tube otorrhea was reported | 94 | 34
  Tube otorrhea was not reported | 35 | 87
Statistical Analysis 1: Comparison: Surgical Management vs Non-Surgical Management; Null hypothesis: There is no difference between the two groups regarding the proportion of children for whom tube otorrhea was reported; Test type: Superiority; Risk Ratio (RR) = 2.57, 95% CI 2-sided [1.91 to 3.48] — [estimate comment as in outcome 1, analysis 1]

14. Secondary Outcome: The Distribution of Children With a Penicillin-Nonsusceptible Nasopharyngeal or Throat Isolate At Any Follow-up Visit According to the Colonization Status at Enrollment
Description: Throat specimens were obtained mainly from children older than 24 months of age. The penicillin-nonsusceptible pathogens considered are penicillin-intermediate and penicillin-resistant Streptococcus pneumoniae and ß-lactamase-positive Haemophilus influenzae. Susceptibility to penicillin was defined as follows: susceptible as a minimum inhibitory concentration (MIC) of <0.1 μg/mL; intermediate as an MIC of 0.1 to 1μg/mL; and resistant as an MIC of >1 μg/mL.
Time Frame: Day 1 until Day 786.
Population: Children with a nasopharyngeal or throat culture at enrollment and at least 1 follow-up nasopharyngeal or throat culture
Measure: Count of Participants; unit: Participants
Arm/Group | Surgical Management | Non-Surgical Management
Number analyzed (Participants) | 113 | 113
Participants
  No pathogens at enrollment: number analyzed (Participants) | 37 | 35
  No pathogens at enrollment: Penicillin-nonsusceptible isolate at a follow-up visit | 25 | 24
  No pathogens at enrollment: No penicillin-nonsusceptible isolate at a follow-up visit | 12 | 11
  Positive only for at least 1 penicillin-susceptible pathogen at enrollment: number analyzed (Participants) | 33 | 35
  Positive only for at least 1 penicillin-susceptible pathogen at enrollment: Penicillin-nonsusceptible isolate at a follow-up visit | 22 | 20
  Positive only for at least 1 penicillin-susceptible pathogen at enrollment: No penicillin-nonsusceptible isolate at a follow-up visit | 11 | 15
  Positive for at least 1 penicillin-nonsusceptible pathogen at enrollment: number analyzed (Participants) | 43 | 43
  Positive for at least 1 penicillin-nonsusceptible pathogen at enrollment: Penicillin-nonsusceptible isolate at a follow-up visit | 38 | 34
  Positive for at least 1 penicillin-nonsusceptible pathogen at enrollment: No penicillin-nonsusceptible isolate at a follow-up visit | 5 | 9
Statistical Analysis 1: Comparison: Surgical Management vs Non-Surgical Management; Null hypothesis: There is no difference between the two groups in the proportion of children with no pathogens at enrollment having a penicillin-nonsusceptible nasopharyngeal or throat isolate at some follow-up visit; Test type: Superiority; Risk Ratio (RR) = 0.96, 95% CI 2-sided [0.74 to 1.24] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Surgical Management vs Non-Surgical Management; Null hypothesis: There is no difference between the two groups in the proportion of children positive only for at least 1 penicillin-susceptible pathogen at enrollment having a penicillin-nonsusceptible nasopharyngeal or throat isolate at some follow-up visit; Test type: Superiority; Risk Ratio (RR) = 1.20, 95% CI 2-sided [0.83 to 1.72] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Surgical Management vs Non-Surgical Management; Null hypothesis: There is no difference between the two groups in the proportion of children positive for at least 1 penicillin nonsusceptible pathogen at enrollment having a penicillin-nonsusceptible nasopharyngeal or throat isolate at some follow-up visit; Test type: Superiority; Risk Ratio (RR) = 1.10, 95% CI 2-sided [0.94 to 1.29] — [estimate comment as in outcome 1, analysis 1]

15. Secondary Outcome: The Distribution of Nonsusceptible Nasopharyngeal or Throat Pathogens Recovered at Episodes of AOM
Description: Throat specimens were obtained mainly from children older than 24 months of age. The penicillin-nonsusceptible pathogens considered are penicillin-intermediate and penicillin-resistant Streptococcus pneumoniae (S. pn) and ß-lactamase-positive Haemophilus influenzae (H. flu). Susceptibility to penicillin was defined as follows: susceptible as a minimum inhibitory concentration (MIC) of <0.1 μg/mL; intermediate as an MIC of 0.1 to 1μg/mL; and resistant as an MIC of >1 μg/mL.
Time Frame: Day 1 until Day 786.
Population: The analysis was ITT. The participants are randomized children with at least one episode of AOM at which a nasopharyngeal or throat culture is obtained.
Measure: Count of Units; unit: Episodes of AOM
Units Other Than Participants: Episodes of AOM
Arm/Group | Surgical Management | Non-Surgical Management
Number analyzed (Participants) | 78 | 88
Number analyzed (Episodes of AOM) | 173 | 196
Episodes of AOM
  Any nonsusceptible pathogen (nonsusceptible S. pn and/or Beta-lactamase positive H. flu) | 66 | 64
  No nonsusceptible pathogen | 107 | 132
Statistical Analysis 1: Comparison: Surgical Management vs Non-Surgical Management; Null hypothesis: There is no difference between the two groups in the proportion of episodes of AOM at which a nonsusceptible pathogen is recovered; Test type: Superiority; Risk Ratio (RR) = 1.14, 95% CI 2-sided [0.84 to 1.55] — [estimate comment as in outcome 1, analysis 1]

16. Secondary Outcome: The Distribution of Nonsusceptible Nasopharyngeal or Throat Pathogens Recovered at Routine Non-Illness Visits
Description: Throat specimens were obtained mainly from children older than 24 months of age. The penicillin-nonsusceptible pathogens considered are penicillin-intermediate and penicillin-resistant Streptococcus pneumoniae (S. pm) and ß-lactamase-positive Haemophilus influenzae (H. flu). Susceptibility to penicillin was defined as follows: susceptible as a minimum inhibitory concentration (MIC) of <0.1 μg/mL; intermediate as an MIC of 0.1 to 1μg/mL; and resistant as an MIC of >1 μg/mL.
Time Frame: Day 1 until Day 786.
Population: The analysis was ITT. The participants are randomized children with at least one routine non-illness visit at which a nasopharyngeal or throat culture is obtained.
Measure: Count of Units; unit: Routine non-illness visits
Units Other Than Participants: Routine non-illness visits
Arm/Group | Surgical Management | Non-Surgical Management
Number analyzed (Participants) | 118 | 113
Number analyzed (Routine non-illness visits) | 485 | 447
Routine non-illness visits
  Any nonsusceptible pathogen (nonsusceptible S. pn and/or Beta-lactamase positive H. flu) | 116 | 98
  No nonsusceptible pathogen | 369 | 349
Statistical Analysis 1: Comparison: Surgical Management vs Non-Surgical Management; Null hypothesis: There is no difference between the two groups in the proportion of routine non-illness visits at which a nonsusceptible pathogen is recovered; Test type: Superiority; Risk Ratio (RR) = 1.09, 95% CI 2-sided [0.84 to 1.41] — [estimate comment as in outcome 1, analysis 1]

17. Secondary Outcome: The Distribution of Nonsusceptible Nasopharyngeal or Throat Pathogens Recovered at AOM Episodes Late During the Respiratory Season (April-May)
Description: as for outcome 15
Time Frame: April 1 to May 31, each of the 2 years of follow-up. The mean length of follow-up was 111 days / 3.7 months.
Population: The analysis was ITT. The participants are randomized children with at least one episode of AOM late during the respiratory season (April-May) at which a nasopharyngeal or throat culture is obtained
Measure: Count of Units; unit: Episodes of AOM
Units Other Than Participants: Episodes of AOM
Arm/Group | Surgical Management | Non-Surgical Management
Number analyzed (Participants) | 27 | 37
Number analyzed (Episodes of AOM) | 37 | 43
Episodes of AOM
  Any nonsusceptible pathogen (nonsusceptible S. pn and/or Beta-lactamase positive H. flu) | 16 | 16
  No nonsusceptible pathogen | 21 | 27
Statistical Analysis 1: Comparison: Surgical Management vs Non-Surgical Management; Test type: Superiority — The analysis was ITT. The participants are randomized children with at least one episode of AOM late during the respiratory season at which a nasopharyngeal or throat culture is obtained; Risk Ratio (RR) = 1.16, 95% CI 2-sided [0.69 to 1.95] — [estimate comment as in outcome 2, analysis 1]

18. Secondary Outcome: The Mean Score Representing Parental Satisfaction With Clinical Management
Description: At the end-of-study visit, parents were asked to rate their level of satisfaction with their child's assigned management using a 5-point scale with higher numbers indicating greater satisfaction, specifically 1 = very dissatisfied, 2 = somewhat dissatisfied, 3 = neither satisfied nor dissatisfied, 4 = somewhat satisfied, and 5 = very satisfied.
Time Frame: The end-of-study visit. The mean day for this visit was 726.
Population: The analysis was ITT. The participants are randomized children who completed the study and whose parent rated their level of satisfaction.
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | Surgical Management | Non-Surgical Management
Number analyzed (Participants) | 105 | 96
Score on a scale | 4.64 (0.10) | 4.43 (0.13)
Statistical Analysis 1: Comparison: Surgical Management vs Non-Surgical Management; Null hypothesis: There is no difference between the two groups in the mean parental satisfaction score; Test type: Superiority; Difference of least-squares means = 0.25, 95% CI 2-sided [-0.06 to 0.56] — [estimate comment as in outcome 8, analysis 1]

19. Secondary Outcome: The Distribution of Parent Reports Indicating At Least One Health Care Encounter Since the Previous Study Visit as an Indicator of Medical Resource Use
Description: Health care encounters, indicators of medical resource use, were ascertained from parent reports. At scheduled study visits, every 8 weeks after randomization. and at interim sick study visits, parents were asked about encounters with healthcare providers, including hospitalizations and visits to emergency departments, urgent care, and primary care providers, since the previous study visit.
Time Frame: Day 1 until Day 786.
Population: The analysis was ITT. The participants are randomized children having at least one parent report.
Measure: Count of Units; unit: Number of parent reports
Units Other Than Participants: Number of parent reports
Arm/Group | Surgical Management | Non-Surgical Management
Number analyzed (Participants) | 122 | 119
Number analyzed (Number of parent reports) | 1635 | 1628
Number of parent reports
  Number of reports indicating at least one health care encounter since the previous study visit | 738 | 672
  Number of reports indicating no health care encounter since the previous study visit | 897 | 956
Statistical Analysis 1: Comparison: Surgical Management vs Non-Surgical Management; Null hypothesis: There is no difference between the two groups in the proportion of parent reports indicating at least one health care encounter since the previous study visit; Test type: Superiority; Risk Ratio (RR) = 1.07, 95% CI 2-sided [0.98 to 1.18] — [estimate comment as in outcome 1, analysis 1]

20. Secondary Outcome: The Distribution of Reported Occurrences of a Parent Missing Work Due to Child's Illness, as an Indicator of Non-Medical Resource Use
Description: Occurrences of parent missing work due to child's illness, an indicator of non-medical resource use, was ascertained from parent reports at scheduled study visits, every 8 weeks after randomization, and at interim sick study visits.
Time Frame: Day 1 until Day 786.
Population: The analysis was ITT. The participants are randomized children having at least one parent report.
Measure: Count of Units; unit: Number of parent reports
Units Other Than Participants: Number of parent reports
Arm/Group | Surgical Management | Non-Surgical Management
Number analyzed (Participants) | 122 | 119
Number analyzed (Number of parent reports) | 1635 | 1628
Number of parent reports
  Number of reports indicating a parent missed work due to child's illness | 286 | 256
  Number of reports indicating parent did not miss work due to child's illness | 1317 | 1342
  Number of reports for which the parent did not answer the question | 32 | 30
Statistical Analysis 1: Comparison: Surgical Management vs Non-Surgical Management; Null hypothesis: There is no difference between the two groups in the proportion of parent reports indicating a parent missed work due to child's illness; Test type: Superiority — Reports for which the parent did not answer the question were excluded from the analysis; Risk Ratio (RR) = 1.11, 95% CI 2-sided [0.88 to 1.41] — [estimate comment as in outcome 1, analysis 1]

21. Secondary Outcome: The Distribution of Reported Occurrences of the Need for Special Childcare Arrangements Due to Child's Illness, as an Indicator of Non-Medical Resource Use
Description: Occurrences of the need for special childcare arrangements due to child's illness, an indicator of non-medical resource use, was ascertained from parent reports at scheduled study visits, every 8 weeks after randomization, and at interim sick study visits.
Time Frame: Day 1 until Day 786.
Population: The analysis was ITT. The participants are randomized children having at least one parent report.
Measure: Count of Units; unit: Number of parent reports
Units Other Than Participants: Number of parent reports
Arm/Group | Surgical Management | Non-Surgical Management
Number analyzed (Participants) | 122 | 119
Number analyzed (Number of parent reports) | 1635 | 1628
Number of parent reports
  Number of reports indicating the need for special child care arrangements due to child's illness | 231 | 195
  Number of reports indicating no need for special child care arrangements due to child's illness | 1402 | 1429
  Number of reports for which the parent did not answer the question | 2 | 4
Statistical Analysis 1: Comparison: Surgical Management vs Non-Surgical Management; Null hypothesis: There is no difference between the two groups in the proportion of parent reports indicating the need for special childcare arrangements due to child's illness; Test type: Superiority — Reports indicating the parent did not answer the question were excluded from the analysis; Risk Ratio (RR) = 1.15, 95% CI 2-sided [0.89 to 1.48] — [estimate comment as in outcome 1, analysis 1]

22. Secondary Outcome: The Mean Scores on the 6 Item Quality of Life Survey Questionnaire (OM-6)
Description: The OM-6 is a 6 item quality of life assessment addressing physical suffering, hearing loss, speech impairment, emotional distress, activity limitations and caregiver concerns. Responses are regarded on an ordinal scale ranging from 1 (no problem) to 7 (greatest problem). The average response, i.e., score, for these 6 items is calculated. The overall child's quality of life (QOL) score, also captured on the OM-6, is expressed on an ordinal response scale that ranges from 0 (worst quality of life) to 10 (best quality). A OM-6 is administered to the parent every 16 weeks after randomization and occasionally at sick visits.
Time Frame: Day 1 until Day 786.
Population: The analysis was ITT. The participants are randomized children having at least one parent report.
Measure: Mean (Standard Error); unit: Score on a scale
Units Other Than Participants: Number of parent reports
Arm/Group | Surgical Management | Non-Surgical Management
Number analyzed (Participants) | 119 | 119
Number analyzed (Number of parent reports) | 890 | 830
Score on a scale
  OM-6 survey score | 1.5 (0.03) | 1.55 (0.03)
  OM-6 survey--Children's overall QOL score | 8.45 (0.07) | 8.37 (0.07)
Statistical Analysis 1: Comparison: Surgical Management vs Non-Surgical Management; Null hypothesis: There is no difference between the two groups in the mean OM-6 survey score; Test type: Superiority; Difference of least-square means = -0.05, 95% CI 2-sided [-0.13 to 0.02] — [estimate comment as in outcome 8, analysis 1]
Statistical Analysis 2: Comparison: Surgical Management vs Non-Surgical Management; Null hypothesis: There is no difference between the two groups in the mean OM-6 survey--children's overall QOL score; Test type: Superiority; Difference of least-square means = 0.06, 95% CI 2-sided [-0.13 to 0.24] — [estimate comment as in outcome 8, analysis 1]

23. Secondary Outcome: The Mean Scores on the 6 Item Caregiver Impact Questionnaire (CIQ)
Description: The Caregiver Impact Questionnaire (CIQ) is a 6 item assessment addressing lack of sleep, absence from work or education, canceling of family activities, changing daily activities, feeling nervous and feeling helpless. Each of these responses is expanded to a continuous scale from 0 (no impact on caregiver) to 100 (greatest impact). The average response, i.e., score, for these 6 items is calculated. The overall caregiver's quality of life (QOL) score, also captured on the CIQ, is expressed on a ordinal response scale that ranges from 0 (worst quality of life) to 10 (best quality). The CIQ is administered to the parent every 16 weeks after randomization and occasionally at sick visits.
Time Frame: Day 1 until Day 786.
Population: The analysis was ITT. The participants are randomized children having at least one parent report.
Measure: Mean (Standard Error); unit: Score on a scale
Units Other Than Participants: Number of parent reports
Arm/Group | Surgical Management | Non-Surgical Management
Number analyzed (Participants) | 119 | 119
Number analyzed (Number of parent reports) | 883 | 818
Score on a scale
  Caregiver impact questionnaire score | 10.82 (0.53) | 10.93 (0.55)
  Caregiver impact questionnaire--Caregiver's overall QOL score | 8.55 (0.06) | 8.50 (0.06)
Statistical Analysis 1: Comparison: Surgical Management vs Non-Surgical Management; Null hypothesis: There is no difference between the two groups in the mean caregiver impact questionnaire score; Test type: Superiority; Difference of least-square means = -0.04, 95% CI 2-sided [-1.55 to 1.47] — [estimate comment as in outcome 8, analysis 1]
Statistical Analysis 2: Comparison: Surgical Management vs Non-Surgical Management; Null hypothesis: There is no difference between the two groups in the mean caregiver impact questionnaire--caregiver's overall QOL score; Test type: Superiority; Difference of least-square means = 0.03, 95% CI 2-sided [-0.14 to 0.20] — [estimate comment as in outcome 8, analysis 1]

24. Secondary Outcome: The Total Cost of Management of Recurrent Acute Otitis Media Per Quality Adjusted Life Days (QALDs) as a Measure of Cost-Effectiveness
Description: Total costs in US dollars were calculated by summing costs of lost wages, office visits, medical procedures, hospitalizations, and medications. Total QALDs were calculated by summing daily utility values. A utility value of 1.0 was assumed for days without AOM, otorrhea, or hospitalization. For days where these states were reported, published utility values associated with each state were used. To arrive at the final measure, total costs were divided by total utility values.
Time Frame: Day 1 until Day 786. The mean length of actual follow-up was 662 days / 1.8 years.
Population: The analysis was ITT. The participants are randomized children.
Measure: Number; unit: US dollars per quality adjusted life day
Arm/Group | Surgical Management | Non-Surgical Management
Number analyzed (Participants) | 129 | 121
US dollars per quality adjusted life day | 7.19 | 5.79

25. Secondary Outcome: The Total Cost of Management of Recurrent Acute Otitis Media Per Quality Adjusted Life Days (QALDs) as a Measure of Cost-Effectiveness According to the Estimated Risk of Acute Otitis Media Recurrences at Enrollment
Description: Total costs in US dollars were calculated by summing costs of lost wages, office visits, medical procedures, hospitalizations, and medications. Total QALDs were calculated by summing daily utility values. A utility value of 1.0 was assumed for days without AOM, otorrhea, or hospitalization. For days where these states were reported, published utility values associated with each state were used. To arrive at the final measure, total costs were divided by total utility values. The estimated risk of AOM at enrollment is described under both Baseline Characteristics and Outcome Measure #2.
Time Frame: Day 1 until Day 786. The mean length of actual follow-up was 662 days / 1.8 years.
Population: The analysis was ITT. The participants are randomized children.
Measure: Number; unit: US dollars per quality adjusted life day
Arm/Group | Surgical Management | Non-Surgical Management
Number analyzed (Participants) | 129 | 121
US dollars per quality adjusted life day
  Children considered at low risk of AOM recurrence: number analyzed (Participants) | 63 | 72
  Children considered at low risk of AOM recurrence | 6.25 | 5.70
  Children considered at high risk of AOM recurrence: number analyzed (Participants) | 66 | 49
  Children considered at high risk of AOM recurrence | 8.00 | 5.91

ADVERSE EVENTS:
Time Frame: The occurrence of adverse events (AEs) were recorded from Day 1 (enrollment) through Day 786. Parents were interviewed at each scheduled study visit, at interim illness visits, and at the end-of-study visit to determine if their child had any adverse events since the preceding visit. All recorded AEs were followed to adequate resolution.
Description: Additionally, during periods of antimicrobial therapy for AOM, parents recorded in an electronic memory aid (or a paper memory aid if an electronic memory aid was unavailable) complete information regarding frequency and consistency of bowel movements, diaper rash necessitating administration of topical antifungal therapy, and otorrhea.
Arm/Group | Surgical Management | Non-Surgical Management
All-Cause Mortality (participants affected / at risk) | 0/129 | 0/121
Serious Adverse Events (participants affected / at risk) | 3/129 | 7/121
Other Adverse Events (participants affected / at risk) | 98/129 | 70/121
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Surgical Management (N=129) | Non-Surgical Management (N=121)
Ileocolic intussusception (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastroenteritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Protocol-defined diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) — Protocol-defined diarrhea was the occurrence of at least three watery stools on 1 day or at least two watery stools on 2 consecutive days, resulting in hospitalization
Asthma exacerbation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) — Includes Asthma exacerbation, Status asthmaticus and Acute bronchospasm
Bronchiolitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory insufficiency (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Complex febrile seizure (Nervous system disorders) | 0 (0) | 1 (1)
Dehydration (General disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Surgical Management (N=129) | Non-Surgical Management (N=121)
Protocol-defined Diarrhea (Gastrointestinal disorders) | 21 (43) | 34 (59) — Protocol-defined diarrhea was the occurrence of at least three watery stools on 1 day or at least two watery stools on 2 consecutive days
Diaper dermatitis (Skin and subcutaneous tissue disorders) | 25 (46) | 33 (56) — Diaper dermatitis was defined as dermatitis resulting in topical antifungal treatment.
Tube otorrhea (Ear and labyrinth disorders) | 94 (320) | 34 (119)
Otorrhea, not tube associated (Ear and labyrinth disorders) | 0 (0) | 8 (8)
Refractory tube otorrhea (Ear and labyrinth disorders) | 3 (4) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-13): https://cdn.clinicaltrials.gov/large-docs/25/NCT02567825/Prot_SAP_002.pdf